CLINICAL TRIAL: NCT04504760
Title: Single and Multiple Ascending Dose Study to Assess the Safety, Tolerability and PK of ONO-2910 in Japanese and Caucasian Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ONO-2910-01
Record Dates: First submitted 2020-07-31; First posted 2020-08-07 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ONO-2910 (Part A and B) (Experimental)
  Interventions: Drug: ONO-2910
- Placebo (Part A) (Placebo Comparator)
  Interventions: Drug: Placebo
- ONO-2910 (Part C and D) (Experimental)
  Interventions: Drug: ONO-2910
- Placebo (Part C and D) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ONO-2910 — Single ascending dose of ONO-2910 will be administered orally.
  Arms: ONO-2910 (Part A and B)
Drug: Placebo — Single dose of placebo will be administered orally.
  Arms: Placebo (Part A)
Drug: ONO-2910 — Multiple ascending dose of ONO-2910 will be administered orally.
  Arms: ONO-2910 (Part C and D)
Drug: Placebo — Multiple dose of placebo will be administered orally.
  Arms: Placebo (Part C and D)

SUMMARY:
To investigate safety, tolerability and pharmacokinetics in Japanese and Caucasian subjects when ONO-2910 is administered as single and multiple doses orally.

DETAILED DESCRIPTION:
This study is the First in Human (FIH) study to investigate safety, tolerability and pharmacokinetics in healthy Japanese and Caucasian adult male subjects when ONO-2910 is administered as single and multiple doses orally. Also, the purpose of this study is to evaluate pharmacokinetics of oral single-dose of ONO-2910 in Japanese elderly male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Japanese healthy adult male subjects (Part A and C)
2. Japanese men or women after menopause aged ≥65 years and ≤74 years (Part B)
3. Caucasian healthy adult male subjects (Part D)
4. Age (at the time of informed consent): ≥20 years, ≤ 45 years (Part A, C and D)

Exclusion Criteria:

1. Subjects currently with or with a history of disease
2. Subjects with current or with a history of severe allergy to drugs or foods
3. Subjects with current or with a history of drug or alcohol abuse

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-03-18 (Actual)

PRIMARY OUTCOMES:
Adverse events [Safety and Tolerability] | Up to 13 days
  Number of participants with adverse events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Cmax [Pharmacokinetic] | Up to 10 days
  Assessment of the Cmax of ONO-2910
Tmax [Pharmacokinetic] | Up to 10 days
  Assessment of the Tmax of ONO-2910
AUC24h [Pharmacokinetic] | Up to 10 days
  Assessment of the AUC24h of ONO-2910
AUClast [Pharmacokinetic] | Up to 10 days
  Assessment of the AUClast of ONO-2910
AUCinf [Pharmacokinetic] | Up to 10 days
  Assessment of the AUCinf of ONO-2910
T1/2 [Pharmacokinetic] | Up to 10 days
  Assessment of the T1/2 of ONO-2910
CL/F [Pharmacokinetic] | Up to 10 days
  Assessment of the CL/F of ONO-2910
fe [Pharmacokinetic] | Up to 4 days
  Assessment of the Vss of ONO-2910
CLr [Pharmacokinetic] | Up to 4 days
  Assessment of the CLr of ONO-2910

CONTACTS AND LOCATIONS:
Overall Officials: Masaharu Komeno, Study Director — Ono Pharmaceutical Co. Ltd
Locations (1):
- Tokyo Clinical Site 01, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No